CLINICAL TRIAL: NCT00088179
Title: A Multicenter, Randomized, Double-Blind, Parallel-group, Placebo-Controlled Study of Pexelizumab in Patients Undergoing Coronary Artery Bypass Grafting With Cardiopulmonary Bypass (PRIMO-CABG II)
Brief Title: Pexelizumab in Patients Undergoing Coronary Artery Bypass Grafting With Cardiopulmonary Bypass (PRIMO-CABG II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Procter and Gamble (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003141
Record Dates: First submitted 2004-07-21; First posted 2004-07-23 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease
Keywords: CABG; CPB
MeSH Terms: conditions — Coronary Artery Disease | interventions — pexelizumab

INTERVENTIONS:
Drug: pexelizumab in conjunction with CABG

SUMMARY:
During a heart bypass procedure, a substance called "complement" is activated by the body. This "complement activation" causes an inflammatory response that can lead to side affects such as chest pain, heart attacks, stroke, heart failure, or death. The purpose of this study is to find out if the study drug (pexelizumab), that blocks "complement activation," can reduce such side effects and be given safely to patients requiring the bypass procedure with the use of the heart-lung machine.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age;
* have 2 or more of the following risk factors:

  • diabetes mellitus; • repeat CABG; • the need for urgent intervention, defined according to the ACC/AHA guidelines as being patients who are required to stay in the hospital due to medical factors, but may be scheduled and operated on within a normal scheduling routine, excluding patients who have had an MI within 48 hours of CABG; • female; • history of a neurologic event (cerebrovascular accident, transient ischemic attack or carotid endarterectomy); • history of congestive heart failure (NYHA CHF Class III or IV); • history of 2 MIs, or an MI that occurred greater than 48 hours but less than 4 weeks prior to CABG;
* provide Informed Consent.

Exclusion Criteria:

* requires salvage intervention as defined by the ACC/AHA guidelines 10 as being ongoing cardiopulmonary resuscitation on the way to the operating room;
* has current cardiogenic shock, acute left ventricular rupture, acute septal rupture or acute papillary muscle rupture;
* has any active bacterial or other infection which is clinically significant, in the opinion of the Investigator (e.g. evaluate the evidence based on WBC, temperature, cultures etc. as appropriate for the patient);
* has a known or suspected hereditary complement deficiency;
* has participated in any other investigational drug study or was exposed to an investigational agent or device within 30 days of randomization;
* is receiving, or is planning to receive, any other investigational drug or device, or will participate in any other research study within 30 days of randomization;
* is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000
Dates: Start 2004-07 (Actual); Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Reduction in mortality.
Reduction in MI incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Peter X Adams, MD, Study Director — Alexion Pharmaceuticals, Inc.; Edward Verrier, MD, Study Chair — University of Washington
Locations (187):
- United States (181):
  - Brookwood Medical Center, Birmingham, Alabama
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - Baptist Health Systems Montclair, Birmingham, Alabama
  - Medical Center East Hospital, Birmingham, Alabama
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Arizona Health Sciences Center, Tucson, Arizona
  - University Medical Center, Tucson, Arizona
  - Southern Arizona Veterans Affairs Health Care System, Tucson, Arizona
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Baptist Medical Center, Little Rock, Arkansas
  - Bakersfield Heart Hospital, Bakersfield, California
  - Seaton Medical Center, Daly City, California
  - Palomar Medical Center, Escondido, California
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Los Angeles County-University of Southern California Medical Center, Los Angeles, California
  - University of Southern California University Hospital, Los Angeles, California
  - St. Vincent Medical Center, Los Angeles, California
  - Veterans Administration Greater Los Angeles Healthcare Sysytem, Los Angeles, California
  - Tri City Medical Center, Oceanside, California
  - University of California Irvine Medical Center, Orange, California
  - Veterans Administration Palo Alto Healthcare System, Palo Alto, California
  - Huntington Memorial Hospital, Pasadena, California
  - Mercy General Hospital, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian St.Luke's Medical Center, Denver, Colorado
  - University of Colorado Health Sciences Center, Denver, Colorado
  - St. Vincent's Medical Center, Bridgeport, Connecticut
  - Hospital of Saint Raphael, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - John F. Kennedy Medical Center, Atlantis, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - North Ridge Medical Center, Fort Lauderdale, Florida
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Regional Medical Center Bayonet Point, Hudson, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - Memorial Hospital, Jacksonville, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Florida Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Wuesthoff Hospital, Rockledge, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Northside Hospital and Heart Institute, St. Petersburg, Florida
  - University Community Hospital, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Atlanta Veteran's Administration (VA) Medical Center, Decatur, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - St. Joseph's/Candler Health System, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Indiana Ohio Heart, Fort Wayne, Indiana
  - Clarian Health Partners, Inc. Methodist Hospital, Indianapolis, Indiana
  - The Indiana Heart Hospital, Indianapolis, Indiana
  - The Heart Center of Indiana, Indianapolis, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - Olathe Medical Center, Olathe, Kansas
  - Galichia Heart Hospital, Wichita, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Veterans Affairs Medical Center, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Terrebonne General Medical Center, Houma, Louisiana
  - Louisiana Heart Hospital, Lacombe, Louisiana
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Oschner Clinic Foundation, New Orleans, Louisiana
  - Pendleton Memorial Methodist Hospital, New Orleans, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - Slidell Memorial Hospital, Slidell, Louisiana
  - Maine Medical Center, Portland, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Union Memorial Hospital, Baltimore, Maryland
  - Peninusla Medical Center, Salisbury, Maryland
  - St. Joseph Medical Center, Towson, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Veterans Administration (VA) Boston Healthcare System, West Roxbury, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - McLaren Regional Medical Center, Flint, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Ingham Regional Medical Center, Lansing, Michigan
  - West Shore Cardiology Research Department, Muskegon, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Covenant Medical Center, Saginaw, Michigan
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - St. Luke's Health System, Kansas City, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Saint Louis University, St Louis, Missouri
  - Des Peres Hospital, St Louis, Missouri
  - Nebraska Heart Hospital, Lincoln, Nebraska
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Cooper Health System/University Medical Center, Camden, New Jersey
  - Our Lady Of Lourdes Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Maimondes Medical Center, Brooklyn, New York
  - United Health Services Hospital, Johnson City, New York
  - New York Presbyterian Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina at Chapel Hill Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - Medcenter One, Bismarck, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals Health System, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - The Dayton Heart Hospital, Dayton, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Good Samaritan Hospital, Zanesville, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - St. Charles Medical Center, Bend, Oregon
  - Legacy Good Samaritan Hospital, Portland, Oregon
  - Doylestown Hospital, Doylestown, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Crozer Chester Medical Center, Upland, Pennsylvania
  - The Chester County Hospital, West Chester, Pennsylvania
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - The Chattanooga Heart Institute, Chattanooga, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Baptist Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Methodist Medical Center, Oak Ridge, Tennessee
  - Heart Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Christus Saint Joseph Hospital, Houston, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - St. Luke's Episcopal Hospital - Texas Heart, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Covenant Medical Center, Lubbock, Texas
  - TexSan Heart Hospital, San Antonio, Texas
  - Northeast Baptist Hospital, San Antonio, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Virginia Hospital Center, Arlington, Virginia
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Memorial Regional Medical Center, Mechanicsville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - CJW Medical Center, Richmond, Virginia
  - Henrico Doctors' Hospital, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- France (4):
  - Hopital Minjoz, Besançon
  - Hopital du Bocage, Dijon
  - Hopital Albert Michallon, Grenoble
  - Hopital Europeen Georges Pompidou, Paris
- Zentrum fuer Herzchirurgie der Frederick-Alexander-Universitaet, Erlangen, Germany
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Smith PK, Shernan SK, Chen JC, Carrier M, Verrier ED, Adams PX, Todaro TG, Muhlbaier LH, Levy JH; PRIMO-CABG II Investigators. Effects of C5 complement inhibitor pexelizumab on outcome in high-risk coronary artery bypass grafting: combined results from the PRIMO-CABG I and II trials. J Thorac Cardiovasc Surg. 2011 Jul;142(1):89-98. doi: 10.1016/j.jtcvs.2010.08.035. Epub 2010 Sep 28. PMID 20880552